CLINICAL TRIAL: NCT00144885
Title: Resonance Magnetic Imaging at the Acute Phase of Endocarditis: Diagnostic and Therapeutic Impact
Brief Title: IMAGE-Endocarditis: Resonance Magnetic Imaging at the Acute Phase of Endocarditis
Acronym: IMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Zakia IDIR, Department Clinical Research of Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: P040431
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2005-09

CONDITIONS: Endocarditis, Bacterial
Keywords: Endocarditis; RMI; Impact measure
MeSH Terms: conditions — Endocarditis, Bacterial; Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (No Intervention)
  Interventions: Behavioral: Modification of therapy

INTERVENTIONS:
Behavioral: Modification of therapy — Modification of the surgery date if adapted, modification of the antibiotics if adapted, based on RMI results

SUMMARY:
Patients with definite or possible infective endocarditis are included in this protocol, at the acute phase of the disease.

DETAILED DESCRIPTION:
Patients with definite or possible infective endocarditis are included in this protocol, at the acute phase of the disease.

Resonance magnetic imaging (head and abdomen) will be performed systematically before Day 7.

The impact on the diagnosis and therapeutic options will be assessed, as compared to pre resonance magnetic nuclear (RMN) imaging declaration.

ELIGIBILITY:
Inclusion Criteria:

* Acute phase of infective endocarditis

Exclusion Criteria:

* Contra indication to RMN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Modification of therapeutic project | As soon as RMI is performed

SECONDARY OUTCOMES:
Modification of diagnostic classification (Duke modified criteria) | As soon as RMI is performed

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Duval, Principal Investigator — Hôpital Bichat, Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital Bichat Claude Bernard, 46 rue Henri Huchard, Paris, France

REFERENCES:
- [Derived] Mahr A, Batteux F, Tubiana S, Goulvestre C, Wolff M, Papo T, Vrtovsnik F, Klein I, Iung B, Duval X; IMAGE Study Group. Brief report: prevalence of antineutrophil cytoplasmic antibodies in infective endocarditis. Arthritis Rheumatol. 2014 Jun;66(6):1672-7. doi: 10.1002/art.38389. PMID 24497495
- [Derived] Iung B, Tubiana S, Klein I, Messika-Zeitoun D, Brochet E, Lepage L, Al-Attar N, Ruimy R, Leport C, Wolff M, Duval X; ECHO-IMAGE Study Group. Determinants of cerebral lesions in endocarditis on systematic cerebral magnetic resonance imaging: a prospective study. Stroke. 2013 Nov;44(11):3056-62. doi: 10.1161/STROKEAHA.113.001470. Epub 2013 Sep 3. PMID 24003046
- [Derived] Iung B, Klein I, Mourvillier B, Olivot JM, Detaint D, Longuet P, Ruimy R, Fourchy D, Laurichesse JJ, Laissy JP, Escoubet B, Duval X; Study Group. Respective effects of early cerebral and abdominal magnetic resonance imaging on clinical decisions in infective endocarditis. Eur Heart J Cardiovasc Imaging. 2012 Aug;13(8):703-10. doi: 10.1093/ehjci/jes023. Epub 2012 Feb 14. PMID 22334638
- [Derived] Duval X, Iung B, Klein I, Brochet E, Thabut G, Arnoult F, Lepage L, Laissy JP, Wolff M, Leport C; IMAGE (Resonance Magnetic Imaging at the Acute Phase of Endocarditis) Study Group. Effect of early cerebral magnetic resonance imaging on clinical decisions in infective endocarditis: a prospective study. Ann Intern Med. 2010 Apr 20;152(8):497-504, W175. doi: 10.7326/0003-4819-152-8-201004200-00006. PMID 20404380